CLINICAL TRIAL: NCT02679677
Title: Evaluation of the Effects of Whole Body Vibration Training With the Galileo Training Device on the Lung Function of Patients With Stable COPD
Brief Title: Evaluation of the Effects of Whole Body Vibration on the Lung Function of Patients With Stable COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: National Center for Tumor Diseases, Heidelberg (Other)
Responsible Party: Principal Investigator, Felix JF Herth, Medical Director, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-607/2014
Record Dates: First submitted 2016-01-18; First posted 2016-02-10 (Estimated); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: COPD
Keywords: Chronic obstructive pulmonary disease; Randomized controlled trial; Physical activity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Sham Comparator): Whole body vibration training as sham procedure (5Hz) 3 times a week, 3x2 minutes, for 6 weeks.
  Interventions: Device: Whole Body Vibration
- Intervention (Experimental): Whole body vibration training (12 Hz up to 30 Hz) 3 times a week, 3x2 minutes, for 6 weeks.
  Interventions: Device: Whole Body Vibration

INTERVENTIONS:
Device: Whole Body Vibration — The principle of the Galileo vibration platform is a side alternating motion similar to a childrens seesaw. Both the amplitude of movement and the frequency of movement may be altered. Frequency may be controlled on the device and settings range from 5Hz to 30Hz. Amplitude of movement is set by spreading one's legs further apart from the midline. Control arm participants remain fixed at 5Hz through the 6 week training period, while intervention arm participants steadily increase their frequency to a maximum of 28Hz.
  Other Names: Galileo; Galileo Platform Novotec Medical

SUMMARY:
The typical clinical progression of COPD usually results in a decreased level of tolerable physical exertion for the patient. The avoidance of strenuous physical activity leads to a deteriorating level of physical fitness, which further decreases the patient's ability to undertake physical activities. Recent research has shown that whole body vibration has the potential to improve physical fitness of participants, including such measures as the 6 minute walking distance. However, information concerning lung function is lacking.

The goal of the study is to test whether the use of whole body vibration training has an effect on the lung function of patients with stable COPD, or if the previously observed effects can be attributed to either pharmaceutical therapy or physical therapy interventions.

ELIGIBILITY:
Inclusion Criteria:

* Stable COPD (Gold II-IV)
* Signed understanding of participation
* The patients must be able to understand and follow the requirements of participation (Understanding of the German language)

Exclusion Criteria:

* Acute thrombosis
* Hemoptysis
* Implants in the targeted training regions (joint implants)
* Acute joint inflammation, active arthrosis or arthropathy.
* Rheumatoid arthritis
* Acute tendinopathy in the targeted training regions
* Acute hernia
* Acute discopathy
* Fresh fracture in the targeted training regions
* Gall or kidney stones
* Wounds still in the process of healing
* Epilepsy
* Severe neurologic disorders (apoplexy, paralysis of upper and lower extremities)
* Severe circulatory disorders (Cardiac insufficiency NYHA > or = III, myocardial infarct less than one month prior, circulatory relevant rhythm disorders, idiopathic syncope)
* Tension pneumothorax
* Acute internal bleeding
* Current therapy with fluoroquinolone
* Alcohol/drug/medication abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
FEV1 | Baseline (T0), Change from baseline measured at end of six weeks of training (T1), Change from baseline measured at six week follow-up measurement (T2)

SECONDARY OUTCOMES:
SGRQ-C: Saint George´s Respiratory Questionnaire for COPD Patients | Baseline (T0), Change from baseline measured at end of six weeks of training (T1), Change from baseline measured at six week follow-up measurement (T2)
mMRC: Modified British Medical Research Council | Baseline (T0), Change from baseline measured at end of six weeks of training (T1), Change from baseline measured at six week follow-up measurement (T2)
CAT: COPD Assessment Test | Baseline (T0), Change from baseline measured at end of six weeks of training (T1), Change from baseline measured at six week follow-up measurement (T2)
PHQ-9 (Brief Patient Health Questionnaire | Baseline (T0), Change from baseline measured at end of six weeks of training (T1), Change from baseline measured at six week follow-up measurement (T2)
SF-12: Short Form (12) Health Questionnaire | Baseline (T0), Change from baseline measured at end of six weeks of training (T1), Change from baseline measured at six week follow-up measurement (T2)
6 Minute Walking Test | Baseline (T0), Change from baseline measured at end of six weeks of training (T1), Change from baseline measured at six week follow-up measurement (T2)
Chair Rising Test | Baseline (T0), Change from baseline measured at end of six weeks of training (T1), Change from baseline measured at six week follow-up measurement (T2)
Handheld Dynamometry Strength Testing of Extremities | Baseline (T0), Change from baseline measured at end of six weeks of training (T1), Change from baseline measured at six week follow-up measurement (T2)
Diffusion capacity for oxygen | Baseline (T0), Change from baseline measured at end of six weeks of training (T1), Change from baseline measured at six week follow-up measurement (T2)
Maximal inspiratory pressure | Baseline (T0), Change from baseline measured at end of six weeks of training (T1), Change from baseline measured at six week follow-up measurement (T2)

CONTACTS AND LOCATIONS:
Overall Officials: Felix Herth, Prof. Dr. med., Principal Investigator — University Hospital Heidelberg
Locations (2):
- Germany (2):
  - Thoraxklinik at Heidelberg University Hospital, Heidelberg
  - University Clinic Gießen and Marburg GmbH, Marburg Campus, Marburg

IPD SHARING:
Plan to Share IPD: Yes